CLINICAL TRIAL: NCT03603288
Title: A Phase III Open-Label Extension Study to Assess the Long-Term Safety and Efficacy of Idebenone in Patients With Duchenne Muscular Dystrophy (DMD) Who Completed the SIDEROS Study
Brief Title: Phase III Study With Idebenone in Patients With Duchenne Muscular Dystrophy (SIDEROS-E)
Acronym: SIDEROS-E
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis concluded to futility of main study SIDEROS (SNT-III-012)
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNT-III-012-E
Expanded Access: NCT03433807 (No longer available)
Record Dates: First submitted 2018-05-31; First posted 2018-07-27 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: respiratory function in DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — idebenone

STUDY DESIGN:
Intervention Model Description: Open-Label Extension Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- idebenone 150 mg film-coated tablets (Experimental): 900 mg idebenone/day (2 tablets to be taken 3 times a day with meal)
  Interventions: Drug: idebenone 150 mg film-coated tablets

INTERVENTIONS:
Drug: idebenone 150 mg film-coated tablets — 900 mg idebenone/day

SUMMARY:
The purpose of the study is to assess the long-term safety and efficacy of idebenone in patients with Duchenne muscular dystrophy (DMD) who completed the SIDEROS study.

DETAILED DESCRIPTION:
The study is an open-label, single-group, multi-center extension study in patients with DMD receiving glucocorticoid steroids who participated in the SIDEROS study and who meet all the inclusion criteria and none of the exclusion criteria for this extension study.

The study consists of 4 study visits scheduled every 6 months (Visit 1/Baseline, Visit 2/Week 26, Visit 3/ Week 52 and Visit 4/ Week 78), and a follow-up visit 4 weeks after treatment discontinuation. Visit 8/Week 78 in SIDEROS study is also SIDEROS-E Visit 1/Baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the SIDEROS study at Visit 8/ Week 78
2. Signed and dated Informed Consent Form for SIDEROS-E

Exclusion Criteria:

1. Patients who discontinued SIDEROS study prematurely (i.e. did not attend all visits from V1 to V8)
2. Safety, tolerability or other issues arising during the course of the SIDEROS study which in the opinion of the Investigator may put the patient at significant risk or may interfere significantly with the patient's participation in the SIDEROS-E study
3. Use of any investigational drug other than the study medication

Min Age: 11 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events, as per ICH Topic E2A | From baseline until visit 4 (week 78)
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Incidence and severity of adverse events, as per ICH Topic E2A | 4 weeks after discontinuation of treatment
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Number of patients with premature discontinuations of study treatment due to adverse events. | From baseline until visit 4 (week 78)
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Number of patients with abnormal safety laboratory parameters. | From baseline until visit 4 (week 78)
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Number of patients with abnormal safety laboratory parameters. | 4 weeks after discontinuation of treatment
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Number of patients with abnormal vital signs. | From baseline until visit 4 (week 78)
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Number of patients with abnormal vital signs. | 4 weeks after discontinuation of treatment
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.
Number of patients with abnormal ECG. | From baseline until visit 4 (week 78)
  To assess the long-term safety of idebenone in DMD patients who completed the SIDEROS study.

SECONDARY OUTCOMES:
Change from Baseline in Forced Vital Capacity (FVC) as percent of predicted (FVC%p). | From baseline until visit 4 (week 78)
  To describe the long-term evolution of respiratory function in idebenone-treated DMD patients who completed the SIDEROS study.
Change from Baseline in Peak Expiratory Flow (PEF) as percent of predicted (PEF%p) | From baseline until visit 4 (week 78)
  To describe the long-term evolution of respiratory function in idebenone-treated DMD patients who completed the SIDEROS study.
Change from Baseline in Forced Expiratory Volume in 1 second (FEV1) as percent of predicted (FEV1%p) | From baseline until visit 4 (week 78)
  To describe the long-term evolution of respiratory function in idebenone-treated DMD patients who completed the SIDEROS study.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (13):
  - University of Alabama - Birmingham, Child Health Research, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - UC Davis Department of Physical Medicine and Rehabilitation, Sacramento, California
  - Center for Integrative Rare Disease Research, Rare Disease Research, LLC, Atlanta, Georgia
  - University of Iowa, Department of Pediatrics, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital Boston, Harvard Medical School, Department of Neurology, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Neurosciences Institute, Neurology - Charlotte Carolinas Healthcare System, Charlotte, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Division of Pulmonology, Philadelphia, Pennsylvania
- Gottfried von Preyer'sches Kinderspital, Vienna, Austria
- Belgium (2):
  - University Hospital Leuven, Leuven
  - CHR Citadelle, Liège
- France (5):
  - Service de neuropédiatrie Pôle Pédiatrie CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Département de pédiatrie - neuropédiatrie, Montpellier
  - Hôpital Hôtel Dieu, Service Explorations Fonctionnelles - Centre de Référence de Maladies Neuromusculaires rares, Nantes
  - I-Motion - Plateforme d'essais cliniques pédiatriques Hôpital Armand Trousseau bâtiment Lemariey porte 20, 2ème étage, Paris
  - Hôpital des enfants, Pédiatrie Neurologie et infectiologie Pôle enfants, Toulouse
- Germany (2):
  - University Medical Center Hamburg - Eppendorf, Department of Paediatrics, Hamburg
  - Center for neuromuscular disorders, Dr. v. Haunersche Kinderklinik, Universität München, München
- Italy (8):
  - Fondazione IRCCS Eugenio Medea, Bosisio Parini
  - U.O. Malattie Neuromuscolari, Istituto Giannina Gaslini, Genova
  - Scientific Coordinator Nemo Sud Clinical CenterAOU Policlinico "G. Martino", Messina
  - Centro Clinico NEMO (NEuroMuscular Omnicentre), Niguarda Hospital, Milan
  - Servizio di Cardiomiologia e Genetica Medica AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - Reparto Di Neurologia dell'Osperdale Di Padova, Padua
  - Dipartimento di Clinica Neurologica e Psichiatrica dell'Eta Evolutiva della Fondazione IRCCS "C. Mondino" di Pavia, Pavia
  - U.O.C. Neuropsichiatria Infantile, Roma
- Spain (2):
  - Hospital Sant Joan de Deu Neuropediatra, Unidad de patologia nueromuscular, Servicio de Neurologia, Barcelona
  - Hospital La Fe de Valencia Avinguda de Fernando Abril Martorell Servicio de Neurologia Torre D, Valencia
- Center for neuromuscular disorders, Universitäts-Kinderspital beider Basel (UKBB), Basel, Switzerland
- United Kingdom (5):
  - Leeds Teaching Hospital NHS Trust, Leeds
  - UCL, National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital for Children, London
  - Clinical Research Facility Level 6 Leazes Wing Royal Victoria Infirmary, Newcastle upon Tyne
  - Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry

REFERENCES:
- [Background] Buyse GM, Voit T, Schara U, Straathof CSM, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, McDonald CM, Rummey C, Meier T; DELOS Study Group. Efficacy of idebenone on respiratory function in patients with Duchenne muscular dystrophy not using glucocorticoids (DELOS): a double-blind randomised placebo-controlled phase 3 trial. Lancet. 2015 May 2;385(9979):1748-1757. doi: 10.1016/S0140-6736(15)60025-3. Epub 2015 Apr 20. PMID 25907158
- [Background] McDonald CM, Meier T, Voit T, Schara U, Straathof CS, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, Rummey C, Leinonen M, Spagnolo P, Buyse GM; DELOS Study Group. Idebenone reduces respiratory complications in patients with Duchenne muscular dystrophy. Neuromuscul Disord. 2016 Aug;26(8):473-80. doi: 10.1016/j.nmd.2016.05.008. Epub 2016 May 12. PMID 27238057
- [Background] Buyse GM, Voit T, Schara U, Straathof CS, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, Rummey C, Leinonen M, Mayer OH, Spagnolo P, Meier T, McDonald CM; DELOS Study Group. Treatment effect of idebenone on inspiratory function in patients with Duchenne muscular dystrophy. Pediatr Pulmonol. 2017 Apr;52(4):508-515. doi: 10.1002/ppul.23547. Epub 2016 Aug 29. PMID 27571420
- [Background] Mayer OH, Leinonen M, Rummey C, Meier T, Buyse GM; DELOS Study Group. Efficacy of Idebenone to Preserve Respiratory Function above Clinically Meaningful Thresholds for Forced Vital Capacity (FVC) in Patients with Duchenne Muscular Dystrophy. J Neuromuscul Dis. 2017;4(3):189-198. doi: 10.3233/JND-170245. PMID 28869486
- See also: SIDEROS study clinicaltrials.gov entry — https://www.clinicaltrials.gov/ct2/show/NCT02814019?term=SIDEROS&rank=1